CLINICAL TRIAL: NCT01911130
Title: Longitudinal Study Comparing the Responsiveness of Outcomes Measures in ALS Trials
Brief Title: Longitudinal Study of Outcomes Measures in ALS Trials
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Patricia L. Andres, Senior Research Scientist, Massachusetts General Hospital
Other Study IDs: 2013P000702
Record Dates: First submitted 2013-07-10; First posted 2013-07-30 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2015-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: outcomes measures; strength measurement; disease progression
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A new strength measurement device called Accurate Test of Limb Isometric Strength (ATLIS) was developed to precisely and conveniently measure static limb strength in patients with ALS. The investigators will compare ATLIS data with data from two commonly used ALS outcomes measures, the ALS Functional Rating Scale-Revised (ALSFRS-R) and slow vital capacity (SVC) in a prospective, longitudinal study. All three outcomes measures will be performed on 100 subjects collected preferably at bi-monthly clinic visits during the study period.

DETAILED DESCRIPTION:
Four sites will participate in data collection for this study and will enroll approximately 20-30 subjects per site. Subjects will be tested every 1 to 4 months for up to two years. Subjects will be tested at each visit using ATLIS, ALSFRS-R questionnaire and slow vital capacity testing.

Inclusion criteria:

* Subjects 18 years or older diagnosed with clinically possible, laboratory supported probable, probable or clinically definite ALS according to the World Federation of Neurology Revised El Escorial Criteria.
* Capable of providing informed consent and complying with trial procedures.

Exclusion criteria:

- Patients, judged by the site clinical investigator to have medical conditions that may limit their ability to safely exert maximal force using the muscles in their arms and legs will be excluded from this study (e.g. unstable hypertension, significant cardiac disease, significant musculoskeletal disorders, or other medical conditions).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* clinically possible, laboartory supported probable, probable or clinically definite ALS according to El Escorial Criteria
* capable of providing informed consent

Exclusion Criteria:

* persons with medical conditions that would limit their ability to safely exert maximal force using muscles in their arms and legs (e.g. unstable cardiac, musculoskeletal, or other medical conditions)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ALS
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Accurate Test of Limb Isometric Strength (ATLIS) between each visit | every 1 to 4 months for up to two years
  ATLIS measures isometric strength in 12 muscle groups in the arms and legs. The subject is tested seated in a specially designed chairs with adjustable uprights. The subject's limb is placed in a standard position and maximal force is exerted on the wireless load cell fixed to the upright. Strength data is digitally captured and expressed as a percentage of expected normal.

SECONDARY OUTCOMES:
Change in ALS Functional Rating Scale - Revised (ALSFRS-R) between each visit | every 1 to 4 months for up to 2 years
  This questionnaire consists of 12 questions about the subject's ability to function in certain daily activities. Questions are asked in an interview format.
Change in Slow Vital Capacity (SVC) between each visit | Every 1 to 4 months for up to two years
  SVC measures the amount of air you can exhale following a deep breath. For this test, we will ask you to hold a mouthpiece in your mouth, breathe in deeply, and breathe out as much air as you can, up to 5 times.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Andres, DPT, MS, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Hershey Medical Center, Hershey, Pennsylvania